CLINICAL TRIAL: NCT01170533
Title: Effects of PPI Therapy on Clopidogrel-Induced Antiplatelet Effects: A Randomized Study
Brief Title: PPI and Clopidogrel Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: UFJ 2009-2
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Drug Interaction
Keywords: proton pump inhibitor; clopidogrel; platelet function
MeSH Terms: interventions — Omeprazole; Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omeprazole (Active Comparator): prospective, open-label, two-sequence, three-period, randomized crossover study
  Interventions: Drug: omeprazole and pantoprazole
- Pantoprazole (Active Comparator): prospective, open-label, two-sequence, three-period, randomized crossover study
  Interventions: Drug: omeprazole and pantoprazole

INTERVENTIONS:
Drug: omeprazole and pantoprazole — The clopidogrel dose will be a 600mg loading dose followed by a 75mg daily maintenance dose, starting the next day for 7 days. Omeprazole will be used at a daily dose of 40mg and pantoprazole at 80mg.

SUMMARY:
Clopidogrel, in combination with aspirin, is currently the recommended treatment for secondary prevention of ischemic events in high-risk patients and for prevention of coronary artery stent thrombosis. Patients receiving aspirin and clopidogrel are frequently treated with proton pump inhibitors, such as omeprazole or pantoprazole, in order to prevent the risk of gastrointestinal bleeding, accorded to guidelines. An interaction between proton pump inhibitors and clopidogrel has been suggested, which may lead to a decrease of clopidogrel effects. It remains unclear whether this interaction between PPIs and clopidogrel might be a class effect or if this may be affected by timing regimen.

The objectives of this two-phase investigation are:

1. to compare clopidogrel platelet inhibitory effects when taken at the same time versus separated at least 8 hours from omeprazole administration.
2. to compare clopidogrel-induced inhibitory effects when taken at the same time versus staggered at least 8 hours from pantoprazole administration.

DETAILED DESCRIPTION:
Clopidogrel, in combination with aspirin, is currently the recommended treatment for secondary prevention of ischemic events in high-risk patients and for prevention of coronary artery stent thrombosis. Patients receiving aspirin and clopidogrel are frequently treated with proton pump inhibitors, such as omeprazole or pantoprazole, in order to prevent the risk of gastrointestinal bleeding, accorded to guidelines. An interaction between proton pump inhibitors and clopidogrel has been suggested, which may lead to a decrease of clopidogrel effects. It remains unclear whether this interaction between PPIs and clopidogrel might be a class effect or if this may be affected by timing regimen. The objectives of this two-phase investigation are: 1. to compare clopidogrel platelet inhibitory effects when taken at the same time versus separated at least 8 hours from omeprazole administration. 2. to compare clopidogrel-induced inhibitory effects when taken at the same time versus staggered at least 8 hours from pantoprazole administration. The clopidogrel dose will be a 600mg loading dose followed by a 75mg daily maintenance dose, starting the next day for 7 days. Omeprazole will be used at a daily dose of 40mg and pantoprazole at 80mg.

The proposed study will have a prospective, randomized, cross-over design. Subjects are randomized in a 1:1 fashion to take PPI concomitantly (CONC regimen) or staggered by 8-12 hours (STAG regimen) for one-week on a background of clopidogrel therapy. In particular, in the CONC regimen both drugs were taken in the morning, while in the STAG regimen clopidogrel was taken in the morning and omeprazole in the evening. After a 2-4 week washout period, subjects crossed-over treatment regimen. After completing these two treatment phases, subjects underwent another washout period of 2-4 weeks and were treated for 1 week with clopidogrel alone, without receiving omeprazole therapy (CLOP regimen). The sequence with the PPI pantoprazole will have the same prospective, randomized, cross-over design as the omeprazole sequence. A CLOP regimen in the absence of pantoprazole will be collected before entering randomization phase with adequate wash-out period.

Blood sampling for platelet function assessments were performed at all three phases of the study at the following time points: a) baseline, b) 24 hours after LD (before intake of study medication), and c) 7 days (24 hours after the last MD).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged between 18 and 75 years

Exclusion Criteria:

1. Known allergies to clopidogrel or omeprazole.
2. Blood dyscrasia or bleeding diathesis.
3. Recent antiplatelet treatment (< 30 days) with a glycoprotein IIb/IIIa antagonist, thienopyridine (ticlopidine, clopidogrel), cilostazol or dipyridamole.
4. Treatment with other medications that may interfere with the CYP system (ketoconazole, itraconazole, diltiazem, erythromycin, clarithromycin, fluvoxamine, fluoxetine, nefazodone, or sertraline).
5. Platelet count <100x106/microL.
6. Diabetes mellitus
7. History of coronary artery disease, gastrointestinal bleed, gastroesophageal reflux disease (GERD), cerebrovascular event or any active malignancy.
8. Active bleeding or hemodynamic instability.
9. Serum creatinine >2mg/dL.
10. Baseline ALT >2.5 times the upper limit of normal.
11. Pregnant females.
12. Patients taking omeprazole or any H2 antagonist or proton pump inhibitors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

REFERENCES:
- [Result] Ferreiro JL, Ueno M, Capodanno D, Desai B, Dharmashankar K, Darlington A, Charlton RK, Bass TA, Angiolillo DJ. Pharmacodynamic effects of concomitant versus staggered clopidogrel and omeprazole intake: results of a prospective randomized crossover study. Circ Cardiovasc Interv. 2010 Oct;3(5):436-41. doi: 10.1161/CIRCINTERVENTIONS.110.957829. Epub 2010 Sep 21. PMID 20858862
- [Result] Ferreiro JL, Ueno M, Tomasello SD, Capodanno D, Desai B, Dharmashankar K, Seecheran N, Kodali MK, Darlington A, Pham JP, Tello-Montoliu A, Charlton RK, Bass TA, Angiolillo DJ. Pharmacodynamic evaluation of pantoprazole therapy on clopidogrel effects: results of a prospective, randomized, crossover study. Circ Cardiovasc Interv. 2011 Jun;4(3):273-9. doi: 10.1161/CIRCINTERVENTIONS.110.960997. Epub 2011 Apr 26. PMID 21521834

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The proposed study will have a prospective, randomized, cross-over design.
Groups:
- Omeprazole: This was a prospective, open-label, two-sequence, three-period, randomized crossover study conducted in non-medicated healthy male subjects between the ages of 18 and 65 years. Subjects were randomized in a 1:1 fashion to take a PPI (omeprazole) concomitantly (CONC) or staggered (STAG) by 8-12 hours for one-week on a background of clopidogrel therapy. In particular, in the CONC regimen both drugs were taken in the morning, while in the STAG regimen clopidogrel was taken in the morning and the PPI (omeprazole)in the evening. After a 2-4 week washout period, subjects crossed-over treatment regimen. After completing these two treatment phases, subjects underwent another washout period of 2-4 weeks and were treated for 1 week with clopidogrel alone, without receiving PPI therapy (CLOP regimen).
- Pantoprazole: This was a prospective, open-label, two-sequence, three-period, randomized crossover study conducted in non-medicated healthy male subjects between the ages of 18 and 65 years. Subjects were randomized in a 1:1 fashion to take a PPI (pantoprazole) concomitantly (CONC) or staggered (STAG) by 8-12 hours for one-week on a background of clopidogrel therapy. In particular, in the CONC regimen both drugs were taken in the morning, while in the STAG regimen clopidogrel was taken in the morning and the PPI in the evening. After a 2-4 week washout period, subjects crossed-over treatment regimen. After completing these two treatment phases, subjects underwent another washout period of 2-4 weeks and were treated for 1 week with clopidogrel alone, without receiving PPI (pantoprazole) therapy (CLOP regimen).
Period: Omeprazole Cross-over
Arm/Group | Omeprazole | Pantoprazole
Started | 20 | 0
Completed | 20 | 0
Not Completed | 0 | 0
Period: Pantoprazole Cross-over
Arm/Group | Omeprazole | Pantoprazole
Started | 0 | 20 (15 participants continued from omeprazole cross-over; the remaining 5 were new participants)
Completed | 0 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This was a prospective, open-label, two-sequence, three-period, randomized crossover study conducted in non-medicated healthy male subjects between the ages of 18 and 65 years. Subjects were randomized in a 1:1 fashion to take a PPI concomitantly (CONC) or staggered (STAG) by 8-12 hours for one-week on a background of clopidogrel therapy. In particular, in the CONC regimen both drugs were taken in the morning, while in the STAG regimen clopidogrel was taken in the morning and the PPI in the evening. After a 2-4 week washout period, subjects crossed-over treatment regimen. After completing these two treatment phases, subjects underwent another washout period of 2-4 weeks and were treated for 1 week with clopidogrel alone, without receiving PPI therapy (CLOP regimen).
  The PPI could be omeprazole (first phase) or pantoprazole (second phase).
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years]
  Omeprazole cross-over n=20 | 34 (6)
  Pantoprazole cross-over n=20 | 33 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Platelet Function as Assessed by the P2Y12 Reactivity Index
Description: P2Y12 reactivity index which will be assessed by flow cytometry determination of vasodilator-stimulated phosphoprotein (VASP).
Time Frame: 1 week
Population: A sample size of 18 patients was required to be able to detect a 10% absolute difference in PRI between both regimens with 80% power and 2-sided significance level of 0.05, assuming a 15% standard deviation for the difference between regimens.
Measure: Least Squares Mean (Standard Error); unit: Percentage of platelet reactivity index
Groups:
- Omeprazole Concomitant: Participants took omeprazole with clopidogrel concomitantly
- Omeprazole Staggered: Participants took omeprazole with clopidogrel staggered
- Pantoprazole Concomitant: Participants took pantoprazole with clopidogrel concomitantly
- Pantoprazole Staggered: Participants took pantoprazole with clopidogrel staggered
- Clopidogrel Only (Omeprazole Phase); Clopidogrel Only (Pantoprazole Phase): Participants took clopidogrel only
Arm/Group | Omeprazole Concomitant | Omeprazole Staggered | Pantoprazole Concomitant | Pantoprazole Staggered | Clopidogrel Only (Omeprazole Phase) | Clopidogrel Only (Pantoprazole Phase)
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Percentage of platelet reactivity index | 56.1 (3.5) | 61.6 (3.4) | 56 (3.9) | 61 (3.9) | 48.8 (3.4) | 61.0 (3.9)

ADVERSE EVENTS:
Arm/Group | Omeprazole | Pantoprazole
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No